CLINICAL TRIAL: NCT00014885
Title: Bone Lead Levels and College Achievement Scores
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 9006-CP-001
Record Dates: First submitted 2001-04-12; First posted 2001-04-13 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Lead Poisoning
Keywords: Lead exposure; Bone lead; Cognitive function; Academic achievement; Neurobehavior
MeSH Terms: conditions — Lead Poisoning

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This project studies the relationship between lead exposure and academic achievement in college students. Most studies of the neurobehavioral effects of lead have focused on performances at the low end of the distribution. There is evidence that lead affects outcome across the entire distribution. This is a retrospective cohort study of subjects whose cognitive function is adequate to gain admission to college. We will use x-ray fluorescence to measure bone lead concentrations in undergraduate college students and test the hypothesis that achievement scores are related to early lead exposure. Early lead exposure has been shown to have measurable effects on academic performance and neurobehavioral outcomes at 18 years of age. Should an effect be found in this study, the spectrum of lead toxicity would be expanded to include subjects with above average function.

ELIGIBILITY:
Current undergraduate student at the University of Pittsburgh who have taken the Scholastic Aptitude Test (SAT).

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 750
Dates: Start 1998-09; Study Completion 2001-08